CLINICAL TRIAL: NCT00705484
Title: Ulcerative Colitis European Registry: A Prospective, Observational, Non-interventional, Post-Marketing Safety Surveillance Program
Brief Title: European Safety Registry in Ulcerative Colitis (P04808)
Acronym: OPUS
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P04808
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Remicade Group: Participants with no prior exposure to Remicade or who have been treated with Remicade in the past, who at the time of enrollment are scheduled to receive Remicade within 30 days of the Baseline Visit. Participants who have been treated in the past with Remicade must have a Remicade-free interval of no less than 90 days from the date of the next expected infusion.
  Interventions: Biological: infliximab
- Standard Therapy Group: Participants who are scheduled to receive standard therapy (defined as initiation or dose-increase of corticosteroids and/or immunosuppressants) that does not include Remicade. Standard therapy participants must not have previously received Remicade for UC or any other condition.
  Interventions: Drug: Standard Therapy

INTERVENTIONS:
Biological: infliximab — The treating physician will determine the treatment regimen and dose of Remicade.
  Other Names: Remicade; SCH 215596
  Groups: Remicade Group
Drug: Standard Therapy — The standard therapy group will consist of participants receiving a treatment regimen that does not include Remicade. The treatment of each standard therapy participant will be left to the discretion of the treating physician and may change during the course of a participant's participation in the registry.
  Groups: Standard Therapy Group

SUMMARY:
This is a prospective, safety surveillance registry in participants with moderate-to-severe active ulcerative colitis (UC).

DETAILED DESCRIPTION:
This is a prospective, observational, post-marketing safety surveillance registry of UC participants treated with Remicade or another standard therapy. Registry centers are targeted to enroll a total of 2000 participants (1000 Remicade participants and 1000 standard therapy participants) and to follow them for a period of up to 5 years. Participants who started the registry on standard therapy may switch over to Remicade.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, of either sex, and of any race.
* Moderate-to-severe active UC, as defined by assessment by the treating physician.
* Must, within 30 days of Baseline, either:

  * Initiate or have a dose increase of immunosuppressive drug(s), including but not limited to systemic steroids (budesonide is considered a topical steroid), azathioprine (AZA), or methotrexate (participants in this category must be Remicade naïve) or
  * Initiate Remicade. Participants who have been treated in the past with Remicade, but who have discontinued for any reason and who are scheduled to receive Remicade within 30 days of the baseline visit must have a Remicade-free interval of no less than 90 days from the date of the next expected infusion
* Must be willing to give written informed consent and must be able to adhere to the procedural requirements of the registry.
* Must be evaluated for active and inactive (latent) tuberculosis (TB) as suggested by local guidelines or as required by the Remicade label for participants starting Remicade.

Exclusion Criteria:

* Female who is known to be pregnant or nursing.
* Previously treated with any other (investigational) biological drug for UC( other than Remicade) prior to Baseline.
* In a situation or have any condition that, in the opinion of the treating physician, may interfere with their optimal participation in the registry.
* Participating in a blinded trial.

In addition, participants with conditions that are contraindicated in the Remicade Summary of Product Characteristics (SPC) should not be treated with Remicade.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants, ages 18 years and older, with a diagnosis of moderate-to-severe active UC will be eligible to enroll in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 2239 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinicaltrials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Panes J, Lindsay JO, Teich N, Lindgren S, Colombel JF, Cornillie F, Flynn HA, Huyck S, Stryszak P, Yao R, Philip G, Reinisch W. Five-year Safety Data From OPUS, a European Observational Safety Registry for Adults With Ulcerative Colitis Treated With Originator Infliximab [Remicade(R)] or Conventional Therapy. J Crohns Colitis. 2019 Sep 19;13(9):1148-1157. doi: 10.1093/ecco-jcc/jjz048. PMID 30809631

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Therapy Group: Participants who are scheduled to receive standard therapy (defined as initiation or dose-increase of corticosteroids and/or immunosuppressants) that does not include Remicade. Standard therapy participants must not have previously received Remicade for Ulcerative Colitis (UC) or any other condition.
Period: Overall Study
Arm/Group | Remicade Group | Standard Therapy Group
Started | 1059 (Number Enrolled) | 1180 (Number Enrolled)
Follow-up Period | 1059 | 296 (Switched From Standard Therapy to Remicade)
Completed | 677 | 772
Not Completed | 382 | 408
Not completed — Adverse Event | 28 | 27
Not completed — Lost to Follow-up | 169 | 250
Not completed — Withdrawal by Subject | 96 | 72
Not completed — Administrative | 89 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remicade Group | Standard Therapy Group | Total
Number analyzed (Participants) | 1059 | 1180 | 2239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (14.24) | 42.0 (15.44) | 41.2 (14.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 464 | 541 | 1005
  Male | 595 | 639 | 1234

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Within Each of Nine Pre-specified Adverse Event (AE) Categories
Description: The nine AE categories are as follows: 1) Serious infections, including infections listed as Serious AEs, tuberculosis, invasive fungal infections, other opportunistic infections, salmonellosis; 2) Infusion-related reactions including delayed hypersensitivity and anaphylactic reactions, and change in severity of infusion-related reactions over time; 3) Fatalities, analyzed by cause; 4)Worsening or new congestive heart failure; 5) Central and peripheral demyelinating neurological disorders; 6) Hematologic conditions such as idiopathic thrombocytopenic purpura, thrombotic thrombocytopenic purpura, thrombocytopenia, pancytopenia, granulocytopenia, leucopenia, hemolytic anemia, aplastic anemia, and thromboembolic events; 7) Malignancies, especially lymphoma, colorectal cancer, and skin cancer; 8) Autoimmune disorders such as lupus and lupus-like syndromes; 9) Hepatobiliary events including autoimmune hepatitis, primary sclerosing cholangitis, and liver function test abnormalities.
Time Frame: Up to 5 years.
Population: All enrolled participants. The Remicade and Standard Therapy Groups are the number of participants who enrolled at the start of the study (N=2239). The Switched to Remicade group are the subset of participants in the Standard Therapy Group, who switched to Remicade.
Measure: Number; unit: Percentage of participants
Groups:
- Switched to Remicade Group: Participants who started the registry on standard therapy but subsequently switched to Remicade. AEs were counted after the switch to Remicade.
Arm/Group | Remicade Group | Standard Therapy Group | Switched to Remicade Group
Number analyzed (Participants) | 1059 | 1180 | 296
Percentage of participants
  Serious Infection | 9.1 | 3.4 | 10.5
  Infusion-Related Reactions | 13.0 | 0.2 | 8.8
  Congestive Heart Failure | 0.3 | 0.3 | 0.3
  Demyelinating Neurological Disorders | 0.1 | 0.2 | 0.3
  Hematologic Conditions | 4.2 | 2.2 | 4.1
  Lymphoproliferative Disorders/ Malignancies | 3.7 | 2.9 | 1.7
  Autoimmune Disorders | 2.2 | 1.1 | 2.4
  Hepatobiliary Events | 4.4 | 3.6 | 4.1
  Fatalities | 0.8 | 1.3 | 0.3

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: All enrolled participants.The Remicade and Standard Therapy Groups are the number of participants who enrolled at the start of the study (N=2239). The Switched to Remicade group are the subset of participants in the Standard Therapy Group, who switched to Remicade.
Groups:
- Switched to Remicade Group: Participants who started in the Standard Therapy Group but switched over to Remicade. AEs were counted after the switch to Remicade.
Arm/Group | Remicade Group | Standard Therapy Group | Switched to Remicade Group
Serious Adverse Events (participants affected / at risk) | 439/1059 | 294/1180 | 102/296
Other Adverse Events (participants affected / at risk) | 321/1059 | 173/1180 | 70/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Remicade Group (N=1059) | Standard Therapy Group (N=1180) | Switched to Remicade Group (N=296)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 2 (3)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Aortic Valve Incompetence (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (4) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Heart Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 6 (7) | 2 (2)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Prinzmetal Angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Node Dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Meniere's Disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Basedow's Disease (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal Scar (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Endocrine Ophthalmopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 10 (10) | 14 (17) | 5 (5)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anal Fissure (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 6 (6) | 3 (3) | 2 (2)
Anal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorectal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorectal Disorder (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 27 (29) | 15 (16) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 243 (370) | 132 (168) | 47 (62)
Colon Dysplasia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 3 (3) | 0 (0)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 3 (5) | 0 (0) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eosinophilic Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric Atony (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric Polyps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal Dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Polyp Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Haemorrhoids Thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileal Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 9 (10) | 0 (0) | 1 (1)
Inflammatory Bowel Disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Intestinal Dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intra-Abdominal Fluid Collection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Jejunal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large Intestinal Stenosis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mesenteric Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0/0 (0) | 1 (1) | 0 (0)
Oedematous Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal Food Impaction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 9 (9) | 8 (8) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0)
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pouchitis (Gastrointestinal disorders) | 7 (9) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Proctitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 6 (6) | 4 (4) | 0 (0)
Rectal Lesion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Stenosis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Small Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1)
Asthenia (General disorders) | 4 (4) | 1 (1) | 0 (0)
Catheter Site Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 2 (2) | 1 (1)
Drug Ineffective (General disorders) | 1 (1) | 0 (0) | 1 (1)
Drug Intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dysplasia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait Disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
General Physical Health Deterioration (General disorders) | 3 (5) | 1 (1) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired Healing (General disorders) | 1 (1) | 2 (3) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Obstruction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 14 (14) | 2 (4) | 4 (4)
Strangulated Hernia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Surgical Failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Treatment Failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular Stent Restenosis (General disorders) | 0 (0) | 2 (2) | 0 (0)
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0)
Cholangitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis Sclerosing (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 4 (4) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholestasis Of Pregnancy (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis Cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis Toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
Serum Sickness (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abdominal Wall Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess Jaw (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acinetobacter Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 6 (9) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
Arthritis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bartholinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Biliary Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Breast Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Candida Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 5 (5) | 2 (2) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus Colitis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)
Cytomegalovirus Infection (Infections and infestations) | 6 (6) | 1 (2) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (5) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eczema Infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Encephalitis Cytomegalovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterococcal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Escherichia Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gallbladder Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 4 (4) | 1 (1)
Gastroenteritis Clostridial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Salmonella (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Incision Site Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious Mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Keratitis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Listeria Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Meningitis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perineal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pilonidal Cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 15 (18) | 5 (5) | 4 (4)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Escherichia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Proctitis Infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Purulent Discharge (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (3) | 1 (2) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rectal Abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Relapsing Fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Renal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory Moniliasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Retinitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Rotavirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pelvic Abscess (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 3 (3) | 1 (1)
Septic Shock (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Tick-Borne Viral Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tubo-Ovarian Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tularaemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (2) | 0 (0)
Viral Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Wound Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anastomotic Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anastomotic Fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anastomotic Leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decompression Sickness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0)
Intestinal Anastomosis Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2)
Open Globe Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Post Procedural Diarrhoea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative Hernia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Stoma Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma Site Discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stoma Site Inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stomal Hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound Evisceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Biopsy Lymph Gland (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Magnesium Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Parathyroid Hormone Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Clostridium Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Endobronchial Ultrasound (Investigations) | 0 (0) | 1 (1) | 0 (0)
Foetal Heart Rate Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 4 (6)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2) | 0 (0)
Lupus-Like Syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Morphoea (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 0 (0) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Clear Cell Sarcoma Of Soft Tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0)
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases To Large Intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (6) | 0 (0)
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Vaginal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Central Nervous System Lesion (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Cerebellar Infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral Ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Gliosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple Sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Optic Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pyramidal Tract Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Quadriparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 0 (0) | 0 (0)
Delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Foetal Death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage In Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Labour Complication (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Labour Pain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Placenta Praevia Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Acute Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Completed Suicide (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 7 (7) | 1 (1) | 0 (0)
Eating Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental Fatigue (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 3 (3)
Acute Prerenal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder Diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder Neck Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus Bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Calculus Urinary (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 2 (2) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Renal Infarct (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Stress Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureteric Stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urethral Stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Cervical Dysplasia (Reproductive system and breast disorders) | 3 (4) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 (3) | 0 (0) | 0 (0)
Noninfective Oophoritis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Perineal Fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Scrotal Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal Fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Bronchial Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7) | 2 (2)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tonsillar Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lentigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pyoderma Gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Solar Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Colectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Female Sterilisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ileostomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ileostomy Closure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic Stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Circulatory Collapse (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 3 (4) | 3 (3) | 1 (1)
Embolism Arterial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Iliac Artery Occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Intermittent Claudication (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Temporal Arteritis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remicade Group (N=1059) | Standard Therapy Group (N=1180) | Switched to Remicade Group (N=296)
Colitis Ulcerative (Gastrointestinal disorders) | 213 (314) | 145 (207) | 51 (75)
Nasopharyngitis (Infections and infestations) | 64 (79) | 23 (25) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 95 (116) | 24 (28) | 17 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.